CLINICAL TRIAL: NCT02686398
Title: Immunogenicity of a Trivalent Influenza Vaccine in Patients With Chronic Kidney Disease Undergoing Hemodialysis: MF59-adjuvanted Versus Non-adjuvanted Vaccines
Brief Title: Immunogenicity of a Trivalent Influenza Vaccine in Chronic Kidney Disease Patients Undergoing Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Hee Jin Cheong, MD, PhD, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KUGH13170
Record Dates: First submitted 2016-01-25; First posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Influenza; End Stage Renal Failure; Chronic Kidney Disease
Keywords: Influenza Vaccines; MF59 oil emulsion; End Stage Renal Failure on Dialysis
MeSH Terms: conditions — Influenza, Human; Renal Insufficiency, Chronic | interventions — fluad vaccine

ARMS (2):
- Fluad (Active Comparator): 88 CKD patients were vaccinated with Fluad.
  Interventions: Biological: Fluad
- Agrippal (Active Comparator): 86 CKD patients were vaccinated with Agrippal.
  Interventions: Biological: Agrippal

INTERVENTIONS:
Biological: Fluad
  Arms: Fluad
Biological: Agrippal
  Arms: Agrippal

SUMMARY:
During the 2013-2014 influenza season, CKD patients undergoing HD participated in the study. The patients were randomized into two groups (MF59-adjuvanted vaccine group or non-adjuvanted vaccine group) and were immunized with the respective vaccine. Sera were collected prior to vaccination and at 1and 6 months post vaccination. Levels of hemagglutination inhibition (HI) antibodies were measured.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease patients undergoing hemodialysis
* Who have given written informed consent at the time of enrollment

Exclusion Criteria:

* Recipients of influenza vaccine of 2013-2014 season before the study
* History of egg allergy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Seroprotection rate (A/H1N1, A/H3N2, B) | 1 month after vaccination
  the proportion of participants with a HI titer level of ≥1:40
Seroconversion rate (A/H1N1, A/H3N2, B) | Change of titer from pre-vaccination to 1 month after vaccination
  the percentage of subjects with either a pre-vaccination HI titer ≥1:10 and a ≥4-fold increase in 1 month after vaccination HI antibody titer from pre-vaccination or pre-vaccination HI titer <1:10 and a 1 month after vaccination HI titer of ≥1:40
GMT fold change (A/H1N1, A/H3N2, B) | Change of GMT from pre-vaccination to 1 month after vaccination
  GMT ratio of the 1 month after vaccination titer to pre-vaccination titer

SECONDARY OUTCOMES:
Seroprotection rate (A/H1N1, A/H3N2, B) | 6 months after vaccination
  the proportion of participants with a HI titer level of ≥1:40
Seroconversion rate (A/H1N1, A/H3N2, B) | Change of titer from pre-vaccination to 6 months after vaccination
  the percentage of subjects with either a pre-vaccination HI titer ≥1:10 and a ≥4-fold increase in 6 months after vaccination HI antibody titer from pre-vaccination or pre-vaccination HI titer <1:10 and a 6 months after vaccination HI titer of ≥1:40
GMT fold change (A/H1N1, A/H3N2, B) | Change of GMT from pre-vaccination to 6 months after vaccination
  GMT ratio of the 6 months after vaccination titer to pre-vaccination titer

CONTACTS AND LOCATIONS:
Overall Officials: Hee Jin Cheong, MD, PhD, Principal Investigator — Korea University Guro Hospital